CLINICAL TRIAL: NCT04518878
Title: Combination of Fixed Low-dose Eltrombopag and rhTPO for Treatment of Immune Thrombocytopenia
Brief Title: Fixed Low-dose Eltrombopag and rhTPO for Immune Thrombocytopenia (FLOWER)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-PKU019
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Immune Thrombocytopenia
Keywords: corticosteroid-resistant or relapsed ITP; eltrombopag; recombinant human thrombopoietin (rhTPO)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fixed Low-dose Eltrombopag and rhTPO (Experimental): Fixed Low-dose Eltrombopag and rhTPO
  Interventions: Drug: Eltrombopag; Drug: rhTPO

INTERVENTIONS:
Drug: Eltrombopag — Fixed dose of eltrombopag oral 25mg daily
  Other Names: Revolade
Drug: rhTPO — Rh-TPO 300U/kg subcutaneous injection once daily for 7 consecutive days, followed by a tapering dose in maintenance therapy.
  Other Names: TPIAO, tebiao

SUMMARY:
This is a prospective, single-arm study to investigate the efficacy and safety of the combination of fixed low-dose eltrombopag plus recombinant human thrombopoietin (rhTPO) as treatment for corticosteroid-resistant or relapsed immune thrombocytopenia (ITP) patients during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Eltrombopag, a small molecule agonist of thrombopoietin receptor (TPO-RA), was recommended as the subsequent treatment for ITP patients, which also already showed robust efficacy.Recombinant human thrombopoietin (rhTPO) is a full-length glycosylated-TPO produced by Chinese hamster ovary cells, which showed its effectiveness in ITP in a variety of studies.

Both eltrombopag and rhTPO demonstrated good safety in ITP patients. Because of their non-immunosuppressive nature, both of them serve as a reasonable choice during the global COVID-19 pandemic.

Since they increase the number of platelets through different mechanisms, and previous studies demonstrated that they might exert synergic effect. The investigators hypothesized that the combination of these two agents could be a promising option for treatment of corticosteroid-resistant or relapsed ITP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed corticosteroid-resistant or relapsed immune thrombocytopenic purpura (ITP)
2. Subject has signed and provided written informed consent.
3. Fertile patients must use effective contraception during treatment and observational period
4. Negative pregnancy test

Exclusion Criteria:

1. Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL
2. Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an aspartate aminotransaminase or alanine aminotransferase level > 3×upper limit of normal
3. Have a New York Heart Classification III or IV heart disease
4. Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures
5. Have active hepatitis B or hepatitis C infection
6. Have a HIV infection
7. Have active infection requiring antibiotic therapy within 7 days prior to study entry
8. Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug
9. Previous splenectomy
10. Had previous or concomitant malignant disease
11. Not willing to participate in the study.
12. Expected survival of < 2 years
13. Intolerant to murine antibodies
14. Immunosuppressive treatment within the last 2 weeks
15. Connective tissue disease
16. Autoimmune hemolytic anemia
17. Patients currently involved in another clinical trial with evaluation of drug treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Complete response | 6 weeks
  A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L.
Response | 6 weeks
  A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia.
No response | 6 weeks
  No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
Relapses | 6 weeks
  A relapses was defined as platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

SECONDARY OUTCOMES:
Early response | 7 days
  Early response was defined as the attainment of a platelet count ≥ 30 × 10⁹ and at least a doubling of baseline platelet count at 1 week.
Initial response | 1 month
  Initial treatment was defined as the attainment of a platelet count ≥ 30 × 10⁹ and at least a doubling of baseline platelet count at 1 month.
TOR (time to response) | 6 weeks
  The time to achieve platelet count ≥ 30×10^9/L and at least 2-fold increase of the baseline count and absence of bleeding since start of treatment.
DOR (duration of response) | 6 weeks
  The duration of achieve platelet count ≥ 30×10^9/L and at least 2-fold increase of the baseline count and absence of bleeding since start of treatment.
Treatments associated adverse events | 6 weeks
  All patients were assessed for safety every week during the first 8 weeks of treatment, and at 2-week intervals thereafter. Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Reduction in bleeding symptoms | 6 weeks
  Changes of bleeding after treatment. Bleeding was defined in accordance with the WHO bleeding scale (0, no bleeding; 1, petechiae; 2, mild blood loss; 3, gross blood loss; and 4, debilitating blood loss).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No